CLINICAL TRIAL: NCT05031091
Title: Epidemiology of Leprosy in French Guiana
Acronym: EPI-LEPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: EPI-LEPR
Record Dates: First submitted 2021-08-24; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hansen's Disease
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: patients with confirmed leprosy: diagnosed or followed up in French Guiana between the beginning of 2006 and the end of 2022
  Interventions: Other: standardised exposure questionnaire
- Control: patient with a dermatological condition not clinically suspicious of leprosy: Any patient, of any age, consulting for a dermatological pathology not clinically suspicious of leprosy during a dermatological consultation by a practitioner of the Cayenne Hospital
  Interventions: Other: standardised exposure questionnaire

INTERVENTIONS:
Other: standardised exposure questionnaire — A standardised exposure questionnaire will be conducted face to face or by telephone. The search for risk factors for leprosy and in particular direct or indirect contact with armadillos will be explored

SUMMARY:
The main objective of the present study is the genotyping of M. leprae strains found in leprosy patients in French Guiana. The secondary objectives are to investigate the presence of M. lepromatosis in these patients, the molecular research of M. leprae resistance to anti-leprosy antibiotics, the study of risk factors for leprosy in humans in Guyana and in particular direct or indirect contact with armadillos, as well as the determination of phylogenetic links between the M. leprae strains found in French Guiana, and with the regional and world reference strains Epidemiology of leprosy in French Guiana.

DETAILED DESCRIPTION:
Rationale: Leprosy (also known as Hansen's disease) is a chronic infection caused by intracellular mycobacteria, Mycobacterium leprae and Mycobacterium lepromatosis (discovered in 2008), preferentially affecting the skin and peripheral nervous system. The disease in humans is potentially disabling and stigmatising.

The modes of transmission of leprosy are not yet fully understood, although it is generally accepted that the main mode of transmission is human-to-human. Apart from humans, the only other major confirmed animal reservoir of M. leprae is the 9-banded armadillo Dasypus novemcinctus, which is found only in the Americas. Recent studies in the southern United States suggest transmission of M. leprae between D. novemcinctus and humans, where 64% of human cases may be attributable to armadillos. Uncertainties remain regarding the zoonotic nature of the disease outside the US and the precise mode of transmission.

The disease is endemic on the American continent where 92% of new cases come from Brazil. In French Guiana - bordering Brazil - leprosy is still present and shows a tendency to recrudesce with about 10 new cases per year. Armadillo consumption is frequent.

Objectives: The main objective of the present study is the genotyping of M. leprae strains found in leprosy patients in French Guiana. The secondary objectives are to investigate the presence of M. lepromatosis in these patients, the molecular research of M. leprae resistance to anti-leprosy antibiotics, the study of risk factors for leprosy in humans in Guyana and in particular direct or indirect contact with armadillos, as well as the determination of phylogenetic links between the M. leprae strains found in French Guiana, and with the regional and world reference strains Population and methods: A cross-sectional study will be conducted on approximately 150 cases of leprosy diagnosed between 2006 and 2022 in French Guyana, seen by the department's anti-leprosy service and for which a skin biopsy (or dermal smear or nasal swab) is available. Genotyping of M. leprae and the search for antibiotic resistance, as well as the search for M. lepromatosis will be carried out by molecular biology. Human strains will be compared with environmental strains from French Guiana and with reference strains found in humans and armadillos. A minimum-spanning-tree and maximum parsimony analysis will be performed to determine the phylogenetic relationships between the different strains.

A 3:1 matched case-control study will be conducted to assess risk factors for leprosy in French Guiana. The 92 cases will be recruited from among leprosy cases diagnosed between 2006 and 2022 in French Guyana, seen by the departmental leprosy control. The 276 controls will be recruited by dermatologists from the Cayenne hospital, throughout the territory, by matching 3 controls per case according to sex and age (± 5 years). A standardised exposure questionnaire will be conducted face to face or by telephone. The search for leprosy risk factors and in particular direct or indirect contact with armadillos (proximity / hunting / handling / consumption) will be explored by univariate and then multivariate conditional logistic regressions taking into account known potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

FOR TRANSVERSAL STUDY:

* any patient, regardless of age, consulting a practitioner at the Cayenne Hospital with a clinical suspicion of leprosy
* Diagnosis of leprosy, confirmed histologically or bacteriologically, made in Guyana between 2006 and 2022
* Skin biopsy (or dermal smear or nasal swab) available in the anatomopathology department of the Andrée Rosemon Hospital and analysable (correct state of preservation and sufficient quantity of tissue)

FOR CASE-CONTROL STUDY - CASES:

* any patient, regardless of age, consulting a practitioner at the Cayenne Hospital with a clinical suspicion of leprosy
* Diagnosis of leprosy, confirmed histologically or bacteriologically, made in Guyana between 2006 and 2022

FOR CASE-CONTROL STUDY - CONTROL:

Any patient, of any age, consulting for a dermatological pathology not clinically suspicious of leprosy during a dermatological consultation by a practitioner of the Cayenne Hospital

Exclusion Criteria:

FOR TRANSVERSAL STUDY:

* Opposition to participation
* Diagnosis of leprosy invalidated after inclusion

FOR CASE-CONTROL STUDY - CASES:

* Opposition to participation
* Inability to answer to the questionnaire
* Diagnosis of leprosy invalidated after inclusion

FOR CASE-CONTROL STUDY - CONTROL:

* Opposition to participation
* Inability to answer to the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For cases: The source population is that of patients with confirmed leprosy, diagnosed or followed up in French Guiana between the beginning of 2006 and the end of 2022, seen in dermatology consultations as part of the Hansen's disease control programme in French Guiana or seen in infectious diseases consultations.
  For controls:The target population for the controls is that of patients with another dermatological pathology in French Guiana. The source population is that of patients seen in consultation by the team of the dermatology department of the Cayenne Hospital for any other reason than leprosy, seen at the Cayenne Hospital or during dermatology consultations carried out in the health centres or at the CHOG.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Genotype of M. Leprae srtrains | 1 day
  Genotyping of M. leprae strains will be genotyped by determining the type (1,2,3,4), subtype (A, B, C, D, E, F, G, H, I, J, K, L, M, N, O, P) by SNP (Single Nucleotide Polymorphism) sequencing and VNTR (Variable Number Tandem Repeat) typing of each selected strain, as recommended by Singh and Cole and used by Truman and Sharma , or, depending on the bacterial index and technical possibilities, by whole genome sequencing, as described by Stefani.

SECONDARY OUTCOMES:
Phylogenetic relationships between strains | 1 day
  Determination of phylogenetic relationships between strains by relative proximity of strains
M. lepromatosis positivity determined by qPCR (real-time PCR) | 1 day
  M. lepromatosis positivity determined by qPCR (real-time PCR)
presence of antibiotic resistance mutation | 1 day
  Presence of antibiotic resistance mutations (primary resistance in samples from new leprosy cases, secondary resistance in samples from retreatment cases (patient diagnosed with leprosy who has already received treatment for leprosy), by PCR or whole genome sequencing
identification of direct contact (hunting/handling/consumption) with armadillos and other wild animals | 1 day
  identification of risk factors for leprosy in humans in French Guiana: Description of the sociodemographic and clinical characteristics of patients
identification of indirect contact (proximity/work on the land) with armadillos and other wild animals | 1 day
  identification of risk factors for leprosy in humans in French Guiana: Description of the sociodemographic and clinical characteristics of patients

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: No